CLINICAL TRIAL: NCT04977726
Title: Resilience Curriculum for Novice Physicians-in-training: a Randomized Controlled, Feasibility Trial.
Brief Title: Resilience Curriculum for Novice Physicians-in-training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University (Other)
Responsible Party: Principal Investigator, Sonja Payne, Assistant Professor, Consultant Anesthesiologist, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11098
Record Dates: First submitted 2021-07-08; First posted 2021-07-27 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRIVE - Simulation Training for Resilience in Various Environments (Experimental)
  Interventions: Behavioral: STRIVE curriculum
- Control (Sham Comparator)
  Interventions: Behavioral: STRIVE curriculum

INTERVENTIONS:
Behavioral: STRIVE curriculum — STRIVE is adapted from the Road to Mental Readiness curriculum, developed by the Department of National Defence in Canada. It is comprised of a 4-hour formal education session where participants are provided knowledge, skills and resources specific to self-assessment for mental wellness and effective mindfulness strategies. High fidelity simulation sessions are then utilized to reinforce and apply mindfulness techniques learned in the formal session.

SUMMARY:
To determine the feasibility of delivering a structured resilience curriculum to novice physicians-in-training, we propose a pilot study to evaluate recruitment rates, course attendance and compliance with follow-up surveys. If our study can demonstrate feasibility in course delivery, further engagement of postgraduate specialty programs will facilitate conduct of an appropriately powered randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All first and second year medical residents enrolled in the Schulich School of Medicine & Dentistry Anesthesia & Emergency Medicine postgraduate residency programs.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Participant Recruitment Potential | 9 months
STRIVE Course Completion | 9 months
  Number of participants randomized to the intervention that complete the STRIVE course
Follow-up Survey Compliance | 9 months

OTHER OUTCOMES:
Self-Reported Resilience at 3 months | 9 months
  Connor-Davidson Resilience Scale (CD-RISC 10). This is a briefer, 10 item version of the full Connor-Davidson Resilience Scale. The scale is 0 to 40 with a higher number representing higher resilience. This scale has been validated in a variety of populations and is a widely used research tool to assess resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No